CLINICAL TRIAL: NCT02219074
Title: A Feasibility Study to Evaluate the Safety and Preliminary Efficacy of the Sebacia Acne Treatment System for the Treatment of Acne Vulgaris
Brief Title: Multiple Arm Study of Sebacia Microparticles in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sebacia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEB-0005
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sebacia microparticle and laser treatment (Experimental)
  Interventions: Device: Sebacia microparticle and laser treatment
- Vehicle and laser treatment (Sham Comparator)
  Interventions: Device: Vehicle and laser treatment

INTERVENTIONS:
Device: Sebacia microparticle and laser treatment
  Arms: Sebacia microparticle and laser treatment
Device: Vehicle and laser treatment
  Arms: Vehicle and laser treatment

SUMMARY:
Prospective, multicenter study with multiple arms to examine the safety and effectiveness of the Sebacia Acne Treatment System for the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of moderate to severe acne vulgaris

Exclusion Criteria:

* use of oral retinoid therapy in the past 12 months
* pregnancy, lactating, or planning to become pregnant
* excessive scarring in the treatment area, or other condition that would impact the ability to evaluate acne

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count | Week 12
Number of adverse events | Screening to 26 weeks

SECONDARY OUTCOMES:
Investigator Global Assessment | Week 12

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Specjalistyczny Gabinet Dermatologiczny, Krakow
  - Military Institute of Health Services, Warsaw